CLINICAL TRIAL: NCT00310011
Title: A Phase II Trial of Gemzar (Gemcitabine), Taxol (Paclitaxel), and Platinol (Cisplatin) (GTP) in Treatment of Advanced Transitional Cell Carcinoma of the Urothelium
Brief Title: Gemcitabine, Paclitaxel, and Cisplatin in Treating Patients With Advanced Cancer of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CCCWFU-88197; CDR0000466059 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-BG98-217; AMGEN-CCCWFU-88197
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; transitional cell carcinoma of the bladder; regional transitional cell cancer of the renal pelvis and ureter; stage IV bladder cancer; recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, paclitaxel, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with paclitaxel and cisplatin works in treating patients with advanced transitional cell cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response to gemcitabine hydrochloride, paclitaxel, and cisplatin (GTP) among patients with regional or distant metastases of transitional cell carcinoma of the urothelium or local/regional recurrence after cystoprostatectomy.
* Determine response in patients who receive GTP as the initial chemotherapeutic treatment as well as in patients who have received prior chemotherapy.
* Determine response duration, freedom from progression, and overall survival.
* Assess the toxicity of GTP.

OUTLINE: This is an open-label study. Patients are stratified according to prior chemotherapy (yes vs no).

Patients receive paclitaxel IV over 3 hours and cisplatin IV over 1 hour on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving a partial response or complete response undergo surgical restaging and debulking. Four to 6 weeks later, patients receive 2 additional courses of chemotherapy.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 71 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma (TCC) of the urothelium (bladder, renal pelvis, or ureter) or TCC with squamous or glandular elements

  * No pure squamous cell carcinoma or adenocarcinoma
* Disease not amenable to local curative treatment
* Regional or distant metastases of TCC of the urothelium OR local/regional recurrence after cystectomy, cystoprostatectomy, nephroureterectomy, or ureterectomy

  * If regional metastases present alone, histological confirmation of the metastases is required
* No clinically evident brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.6 mg/mL
* Bilirubin ≤ 1.8 mg/mL
* SGOT ≤ 3 times upper limit of normal
* Life expectancy > 3 months
* No known sensitivity to E. coli-derived products
* No other prior or concurrent malignancy except active/inactive nonmelanoma skin cancer, adequately treated stage I or II cancer currently in complete remission, or observation-only early-stage prostate cancer
* No other serious medical illness that would limit survival to < 3 months
* No psychiatric condition that would limit compliance with study requirements
* No active uncontrolled bacterial, viral, or fungal infection unless corrected or controlled
* No hemorrhagic disorder
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic chemotherapy regimen
* Prior intravesical therapy allowed
* Prior definitive radiation to renal pelvis, ureter, or bladder allowed
* No concurrent chemotherapy with nonstudy drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 1998-06; Primary Completion 2005-10 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Response
Response duration
Freedom from progression
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Frank M. Torti, MD, MPH, Study Chair — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Regional Cancer Center, Greensboro, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina